CLINICAL TRIAL: NCT07359339
Title: Microneedling With Platelet Rich Plasma Versus Microneedling Alone For Gingival Depigmentation: A Randomized Controlled Clinical Trial
Brief Title: Microneedling With Platelet Rich Plasma Versus Microneedling Alone For Gingival Depigmentation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelrahman Sameer Abdullah, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PER 3_3_1.1
Record Dates: First submitted 2025-12-18; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Gingival Pigmentation
Keywords: Pigmentation; Gingiva; PRP; Microneedling
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microneedling will be done with application of Platelet Rich Plasma for depigmentation. (Experimental): A Dermapen device will be used to microneedle the gingival tissue (model M8) with 24 microneedles arranged in rows, which is adjusted according to the gingival thickness at the 6th mode speed of 700 cycles/min(Mostafa and Alotaibi 2022).
  It will be laid perpendicular to gingival surface and MN will be carried out in horizontal, vertical and diagonal directions about four to five times for the whole hyperpigmented gingiva until mild microbleeding and mild erythema was clearly visible.
  Once bleeding points are observed on all areas of the pigmented gingiva, it will be irrigated using saline solution and dried using sterile gauze.
  Patients receive injection of PRP in their Gingiva. To prepare PRP, 10mL of the patient's venous blood sample was taken manually with a sterile 10mL syringe and then centrifuged with 1300 RPM/10min, buffy coat and plasma were then extracted and re-centrifuged with 2000 RPM/10min. The injection of 1mL of PRP was immediately initiated .
  Interventions: Procedure: Microneedling will be done with application of Platelet Rich Plasma for depigmentation.
- Microneedling will be done alone for Gingival depigmentation. (Active Comparator): A Dermapen device will be used to microneedle the gingival tissue (model M8) with 24 microneedles arranged in rows, which is adjusted according to the gingival thickness at the 6th mode speed of 700 cycles/min(Mostafa and Alotaibi 2022).
  It will be laid perpendicular to gingival surface and MN will be carried out in horizontal, vertical and diagonal directions about four to five times for the whole hyperpigmented gingiva until mild microbleeding and mild erythema was clearly visible.
  Once bleeding points are observed on all areas of the pigmented gingiva, it will be irrigated using saline solution and dried using sterile gauze.
  Interventions: Procedure: Microneedling alone for Gingival Depigmentation.

INTERVENTIONS:
Procedure: Microneedling will be done with application of Platelet Rich Plasma for depigmentation. — A Dermapen device will be used to microneedle the gingival tissue (model M8) with 24 microneedles arranged in rows, which is adjusted according to the gingival thickness at the 6th mode speed of 700 cycles/min(Mostafa and Alotaibi 2022). It will be laid perpendicular to gingival surface and MN will be carried out in horizontal, vertical and diagonal directions about four to five times for the whole hyperpigmented gingiva until mild microbleeding and mild erythema was clearly visible. Once bleeding points are observed on all areas of the pigmented gingiva, it will be irrigated using saline solution and dried using sterile gauze. Patients receive injection of PRP in their Gingiva. To prepare PRP, 10mL of the patient's venous blood sample was taken manually with a sterile 10mL syringe and then centrifuged with 1300 RPM/10min, buffy coat and plasma were then extracted and re-centrifuged with 2000 RPM/10min. The injection of 1mL of PRP was immediately initiated .
  Other Names: PRP
  Arms: Microneedling will be done with application of Platelet Rich Plasma for depigmentation.
Procedure: Microneedling alone for Gingival Depigmentation. — A Dermapen device will be used to microneedle the gingival tissue (model M8) with 24 microneedles arranged in rows, which is adjusted according to the gingival thickness at the 6th mode speed of 700 cycles/min(Mostafa and Alotaibi 2022).
  It will be laid perpendicular to gingival surface and MN will be carried out in horizontal, vertical and diagonal directions about four to five times for the whole hyperpigmented gingiva until mild microbleeding and mild erythema was clearly visible.
  Once bleeding points are observed on all areas of the pigmented gingiva, it will be irrigated using saline solution and dried using sterile gauze.
  Arms: Microneedling will be done alone for Gingival depigmentation.

SUMMARY:
To evaluate the usage of microneedling with platelet rich plasma as a gingival depigmentation method in comparison to microneedling alone for pigment intensity reduction.

Pre-operative preparation phase includes ultrasonic scaling and oral hygiene instructions for all patients. Eligible patients will be randomly allocated into two groups.

Clinical photographs: Clinical photographs will be taken at baseline, 1 and 6 months postoperatively.

Intervention Group (Group A): Microneedling will be done with application of Platelet Rich Plasma for depigmentation.

Control Group (Group B): microneedling will be done alone for depigmentation.

DETAILED DESCRIPTION:
In both groups:

Local anesthesia (Articaine with 1:100,000 Epinephrine( will be administered by infiltration technique).

A Dermapen device will be used to microneedle the gingival tissue (model M8) with 24 microneedles arranged in rows, which is adjusted according to the gingival thickness at the 6th mode speed of 700 cycles/min.

It will be laid perpendicular to gingival surface and MN will be carried out in horizontal, vertical and diagonal directions about four to five times for the whole hyperpigmented gingiva until mild microbleeding and mild erythema was clearly visible.

Once bleeding points are observed on all areas of the pigmented gingiva, it will be irrigated using saline solution and dried using sterile gauze.

Intervention group:

Patients receive injection of PRP in their Gingiva. To prepare PRP, 10mL of the patient's venous blood sample was taken manually with a sterile 10mL syringe and then centrifuged with 1300 RPM /10min, buffy coat and plasma were then extracted and re-centrifuged with 2000 RPM /10min. The injection of 1mL of PRP was immediately initiated with a 1 cc insulin syringe 30G, (0.1mL in each point of injection).

Postoperative Care:

Patients were instructed to refrain from mechanical oral hygiene practices in regard to the target region for the day of the operation following each visit to minimize mechanical damage to the treated areas.

If discomfort or itching was reported on the first day, analgesics were prescribed (Brufen 400 mg tablets, two times daily after meal).

Restricted spicy, acidic, and coloring food. Antiseptic mouth rinse 0,12% chlorhexidine rinse were prescribed, for 60 seconds two times a day for 14 days.

Apply an ice pack to the treated area for the first 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* • Patients exhibiting melanin hyperpigmentation in the anterior region of the upper or lower gingiva.

  * Age ≥ 18 year old.
  * Patients should be free from any systemic diseases according to modified Cornell Medical index (Abramson 1966).
  * Non- smokers

Exclusion Criteria:

* • Fully edentulous patients.

  * Patients with endocrine disorders causing hyperpigmentation or drug induced gingival pigmentation. (Sreeja, Ramakrishnan et al. 2015)
  * Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Dummett-Gupta Oral Pigmentation Index (DOPI) | 6 months
  the degree of gingival pigmentation is scored as 0, pink tissue [no clinical pigmentation]; 1 = mild light brown tissue [mild clinical pigmentation]; 2, medium brown or mixed brown and pink tissue [moderate clinical pigmentation]; or 3, deep brown/blue-black tissue [heavy clinical pigmentation]

SECONDARY OUTCOMES:
Pain (Becker et al., 2018) | 7 days after intervention.
  Using Visual analogue score questionnaire, A number from 0 to 10 ( 10 for the most pain experience and 0 for no pain experience).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo university, Cairo, El Manial
  - Faculity of Dentistry, Cairo university, Cairo, El Manyl

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT07359339/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT07359339/ICF_001.pdf